CLINICAL TRIAL: NCT01729117
Title: The 1,2,3 Plan: A Randomized Controlled Trial of Meal Replacement With a Lifestyle Modification Program vs. Standard Care at a Community Diabetes Clinic Serving a Low Socioeconomic Hispanic Population
Brief Title: A Trial of Meal Replacement at a Community Diabetes Clinic Serving a Low Socioeconomic Hispanic Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-08-00646
Record Dates: First submitted 2012-11-13; First posted 2012-11-20 (Estimated); Last update posted 2012-11-20 (Estimated); Status verified 2012-11

CONDITIONS: Type 2 Diabetes; Obesity
Keywords: Type 2 diabetes; Obesity; Insulin; Hispanic; Low-income; Meal replacement
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Insulin Resistance | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Meal Replacement (Other): Meal Replacements will be provided to participants randomized to the MR group
  Interventions: Other: Meal Replacement
- Standard Care (Other): Standard Care participants will receive standard care but no meal replacements
  Interventions: Other: Standard Care

INTERVENTIONS:
Other: Meal Replacement — 5 Meal Replacements/day will be given for 3 months and then 1/day for 9 months.
  Other Names: HMR70 Plus products; HMR Boston, Massachusetts
  Arms: Meal Replacement
Other: Standard Care — Standard Care only
  Arms: Standard Care

SUMMARY:
Background and Rationale Research studies have shown that patients with type 2 diabetes (T2DM) who lose weight have better glucose control and less risk for heart disease. It has been difficult to achieve these results in a non-research setting. Meal replacements (MR) are pre-packaged meals with appropriate calories and nutrients that enhance adherence to a weight loss program by reducing decision-making and facilitating target caloric intake. The University of Southern California (USC) arm of the NIH funded Look AHEAD study at Roybal Clinic has demonstrated acceptability and success of MRs in conjunction with a structured lifestyle modification program in achieving weight loss in underserved Hispanic T2DM patients.

Objectives Our short-term objective is to determine the efficacy, safety and feasibility of a 3-month full MR program in conjunction with a 1 year standardized lifestyle modification program in a clinic setting. Our longer-term goal is to acquire data for sample size and power estimates for a larger NIH- or other funded prospective, randomized trial.

Study Methodology A 1-year, prospective trial study of 30 obese subjects with T2DM treated with insulin randomized to 2 groups: standard care (SC) or Meal Replacement group (MR). The SC will receive usual care at Roybal Diabetes Management Clinic (DMC). The MR will receive MRs and a lifestyle course in addition to the usual clinical care at the Roybal DMC. Phase 1 consists of 3-months 1200 -1400cal diet using full MR. Phase 2 consists of a 3-month transition to the same caloric intake using regular meals and 1 MR/day . Phase 3 consists of a 6-month weight loss maintenance period with 1 MR/day. This will be about 1400-1600 calories/day for women and 1800 to 2000 calories/day for men. Individual and group educational, support and counseling visits will be components of all 3 phases of the study.

Outcomes Efficacy of the program will be determined by weight, waist measurement and waist to hip ratio, blood pressure, HbA1c, lipids, and medication use at baseline and at 3, 6, 9 and 12 months. These are all measurements that are done routinely in these patients. Safety will be determined by monitoring of adverse events.

Data Analysis We will compare the outcomes between the SC and MR at 0,3,6,9 and 12 months to determine if there is evidence that the intervention improves outcomes and is safe.

ELIGIBILITY:
Inclusion Criteria:

Demographic

* Age >18 years
* Enrolled in the Roybal Diabetes Management Clinic
* Self-described as Hispanic
* Willing and able to participate in Spanish language group sessions.
* Willing and able to attend study visits for the duration of the study at the allocated times.
* Willing and able to maintain a food exercise and medication log and perform and record self-monitoring of blood glucose (SMBG) Clinical
* T2DM diagnosed by fasting blood glucose >126mg/dL or random blood glucose >200mg/dL
* BMI>30 kg/m2
* If a woman of childbearing potential, using effective contraception. Biochemical HbA1c 8%-12% Medication
* On insulin therapy

Exclusion Criteria:

Medical conditions

* Type 1 DM
* Illness likely to lead to unstable weight or altered glucose control.
* Proliferative diabetic retinopathy on eye examination within the last 6 months.
* Gallstones suspected on clinical history or documented on ultrasound.
* Serum creatinine >1.5mg/dL
* Symptomatic cardiovascular disease
* Documented liver disease other than fatty liver
* Lactating, pregnant or intending to become pregnant within the following year Psycho-social conditions
* Inability or unwillingness to participate in a Spanish-language lifestyle group.
* Eating disorder such as bulimia
* Uncontrolled psychiatric disorder such as severe uncontrolled depression or bipolar disorder.
* Inability to attend scheduled appointments regularly for the duration of the study Medication use
* Use of weight loss medication within previous 3 months including exenatide.
* Use of medication (other than diabetes medication) likely to lead to unstable weight or altered glucose control
* Laxative or substance abuse
* More than 10 alcoholic drinks/week

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-05; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Change in BMI | 12months

SECONDARY OUTCOMES:
Severe Hypoglycemic Events | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth O Beale, MD, Principal Investigator — University of Southern California
Locations (1):
- Roybal Diabetes Management Clinic, Los Angeles, California, United States